CLINICAL TRIAL: NCT01071070
Title: A Phase 3b, Randomized, Active-Controlled, Single-Blind, Multicenter Study to Evaluate the Safety and Efficacy of Paricalcitol Injection in Reducing Serum Intact Parathyroid Hormone Levels in Chronic Kidney Disease Stage 5 Subjects Receiving Hemodialysis
Brief Title: Evaluate Safety and Efficacy of Paricalcitol in Reducing Serum Intact Parathyroid Hormone in Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: M06-823
Record Dates: First submitted 2009-11-25; First posted 2010-02-19 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Secondary hyperparathyroidism
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group 1 (Active Comparator): Initial dosing based on a formula of intact parathyroid hormone value/80 (where intact parathyroid hormone value is the baseline value in pg/mL).
  Interventions: Drug: paricalcitol
- Group 2 (Active Comparator): Dose determined by US paricalcitol injection package insert dosing instructions (starting dose at 0.04 microgram/kg)
  Interventions: Drug: paricalcitol

INTERVENTIONS:
Drug: paricalcitol — Initiation dosing based on 2 approved package inserts , followed by a dose adjusted by limited chemistry test value. See Arm Description for additional details.
  Other Names: ABT-358; Zemplar

SUMMARY:
Evaluate Safety and Efficacy of Paricalcitol in Reducing Serum Intact Parathyroid Hormone in Chronic Kidney Disease

DETAILED DESCRIPTION:
Evaluate the safety and efficacy of paricalcitol injection with two different dosing regimens (currently approved dosing regimen used in the US package insert versus dosing based on a formula of iPTH/80 that was approved and used in the EU package insert) in Chronic Kidney Disease (CKD) Stage 5 subjects with secondary hyperparathyroidism receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a Chinese male or female greater than or equal to 20 years old.
2. Subject is diagnosed with Chronic Kidney Disease Stage 5 and must be on maintenance hemodialysis three times a week for at least 2 months prior to the Screening Visit and expected to remain on hemodialysis for the duration of the study.
3. For entry into the Treatment Phase, the subject must have:

   * Intact parathyroid hormone greater than or equal to 300 pg/mL
   * Serum calcium less than 10.2 mg/dL (2.55 mmol/L)
   * Calcium-phosphorus product less than 65 mg^2/dL^2

Exclusion Criteria:

1. Subject has a history of an allergic reaction or significant sensitivity to vitamin D or vitamin D related compounds.
2. Subject received a partial parathyroidectomy within one year prior to the Screening Phase.
3. Subject with New York Heart Association (NYHA) Class III or IV.
4. Subject has taken aluminum-containing phosphate binders for greater than 3 weeks in the last 3 months prior to the Screening Phase, or requires such medications for greater than 3 weeks in the study.
5. Subject has a current malignancy (with the exception of basal or squamous cell carcinoma of the skin), or clinically significant liver disease, in the opinion of the Investigator.
6. Subject has a history of drug or alcohol abuse within 6 months prior to the Screening Phase.
7. Subject is known to be human immunodeficiency virus (HIV) positive.
8. Subject has evidence of poor compliance with diet, medication or hemodialysis that may interfere, in the Investigator's opinion, with adherence to the protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Kang, MD, Study Director — Abbott (China)
Locations (12):
- China (12):
  - Site Reference ID/Investigator# 23483, Beijing
  - Site Reference ID/Investigator# 23485, Beijing
  - Site Reference ID/Investigator# 23482, Beijing
  - Site Reference ID/Investigator# 23484, Dalian
  - Site Reference ID/Investigator# 23486, Guangzhou
  - Site Reference ID/Investigator# 23488, Nanjing
  - Site Reference ID/Investigator# 37722, Qingdao
  - Site Reference ID/Investigator# 23490, Shanghai
  - Site Reference ID/Investigator# 25502, Shanghai
  - Site Reference ID/Investigator# 23489, Shanghai
  - Site Reference ID/Investigator# 23487, Shanghai
  - Site Reference ID/Investigator# 35822, Wenzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at investigative sites in China. Recruitment began in October 2009 and ended in July 2010. The study population consisted of participants with Stage 5 chronic kidney disease who were receiving hemodialysis.
Pre-assignment Details: If subjects were receiving vitamin D receptor (VDR) activators, they participated in a Washout Phase for 2 weeks prior to entering into the Screening Phase in order to wash out any VDR activators and their potential hysteresis or carryover effects.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 108 | 108
Completed | 104 | 105
Not Completed | 4 | 3
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Missed 3 consecutive doses of study drug | 2 | 0
Not completed — Hypercalcemia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 108 | 108 | 216
Age Continuous [Mean (Standard Deviation); unit: years] | 50.5 (13.55) | 50.8 (12.67) | 50.6 (13.09)
Age, Customized [Number; unit: Participants]
  < 65 years | 91 | 93 | 184
  >=65 years | 17 | 15 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 77
  Male | 67 | 72 | 139
Region of Enrollment [Number; unit: participants]
  China | 108 | 108 | 216

OUTCOME MEASURES:

1. Primary Outcome: The Achievement of Two Consecutive Greater Than or Equal to 30% Decreases From Baseline Intact Parathyroid Hormone Levels
Description: The number of participants who achieved (Yes) or did not achieve (No) two consecutive decreases of greater than or equal to 30% from baseline in intact parathyroid hormone (iPTH) values
Time Frame: Baseline to 12 Weeks
Population: The analysis was based on the per-protocol population, which consisted of all randomized participants who completed at least 6 weeks of treatment and met the conditions that defined the per-protocol population.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 105 | 102
participants
  Yes | 93 | 57
  No | 12 | 45

2. Secondary Outcome: The Proportion of Subjects Achieving a Final Intact Parathyroid Hormone Value Between 150 and 300 pg/mL
Description: The number of subjects with (Yes) or without (No) final intact parathyroid hormone (iPTH) values between 150 and 300 pg/mL
Time Frame: Baseline to 12 Weeks
Population: The analysis was based on the intent-to-treat (ITT) population, which consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
participants
  Yes | 19 | 21
  No | 89 | 87

3. Secondary Outcome: The Change From Baseline to the Final Observation in Intact Parathyroid Hormone Value
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
pg/mL | -342.57 (43.82) | -191.53 (43.82)

4. Secondary Outcome: The Change From Baseline to the Final Observation in Calcium
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
mg/dL | 0.64 (0.06) | 0.59 (0.06)

5. Secondary Outcome: The Change From Baseline to the Final Observation in Calcium-phosphorus Product
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg^2/dL^2
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
mg^2/dL^2 | 7.53 (1.47) | 8.15 (1.47)

6. Secondary Outcome: The Change From Baseline to the Final Observation in the Vital Sign of Systolic Blood Pressure
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
mm Hg | -1.47 (19.76) | -1.75 (21.03)

7. Secondary Outcome: The Change From Baseline to the Final Observation in the Vital Sign of Diastolic Blood Pressure
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
mm Hg | -1.47 (11.31) | -0.32 (13.68)

8. Secondary Outcome: The Change From Baseline to the Final Observation in the Vital Sign of Heart Rate
Time Frame: Baseline to 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
beats per minute | 0.51 (9.48) | -0.89 (11.38)

9. Secondary Outcome: The Proportion of Subjects With 2 Consecutive Calcium Measurements Greater Than 11.0 mg/dL (2.75 mmol/L)
Description: The number of subjects with (Yes) or without (No) two consecutive calcium measurements greater than 11.0 mg/dL (2.75 mmol/L)
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 108 | 108
participants
  Yes | 1 | 0
  No | 107 | 108

ADVERSE EVENTS:
Time Frame: From the time of study drug administration until 30 days following discontinuation of study drug administration.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/108 | 3/108
Other Adverse Events (participants affected / at risk) | 29/108 | 19/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=108) | Group 2 (N=108)
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=108) | Group 2 (N=108)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 6
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.